CLINICAL TRIAL: NCT04190953
Title: Skeletal, Dental and Upper Airway Changes in Skeletal Class II Division 1 Patients With the Constricted Maxilla (8-14 Years Old) Treated With Twin Block and Hyrax, Evaluated Through Pressure Drop Experimental Analysis.
Brief Title: Upper Airway's Pressure Drop Analyses After Mandibular Advancement and Maxillary Expansion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00095427
Record Dates: First submitted 2019-11-21; First posted 2019-12-09 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Apnea; Airway Obstruction, Nasal; Mandible Small; Maxillary Hypoplasia
MeSH Terms: conditions — Apnea; Nasal Obstruction; Micrognathism; Retrognathia

STUDY DESIGN:
Intervention Model Description: Twin block and Hyrax appliances will be installed in 1/3 of the patients, while hyrax and twin block devices will be applied to the other 1/3 of the patients. Another 1/3 of patients will be the control group with no treatment
Who Masked: Outcomes Assessor
Masking Description: When data will be analyzed, data will be coded to keep confidentiality for time and type of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Twin Block then Hyrax (Experimental): Patients will undergo mandibular advancement prior to maxillary expansion using Twin block prior to Hyrax
  Interventions: Other: Twin block then Hyrax
- Hyrax then Twin block (Experimental): Patients will undergo maxillary expansion prior to mandibular advancement using Hyrax prior to Twin block
  Interventions: Other: Hyrax then Twin block
- Control (No Intervention): Patients will wait 1,5 years before the start of treatment

INTERVENTIONS:
Other: Twin block then Hyrax — Patients will undergo mandibular advancement prior to maxillary expansion
  Arms: Twin Block then Hyrax
Other: Hyrax then Twin block — Patients will undergo maxillary expansion prior to mandibular advancement
  Arms: Hyrax then Twin block

SUMMARY:
Breathing is a crucial function for everyone. Breathing impairment in children could lead to behavioral and cognitive problems at least. But what if orthodontic treatment could help those patients to breathe better, with less effort? This research proposal aims to find out if the increase in the upper airway volume seen in some research results can be related to a decrease in respiratory effort and an improvement in the breathing capacity of those patients. In other words, if a tube shape is changed or if a tube is enlarged, would the airflow passing inside the tube change in velocity? Or would there be more air? Therefore, investigating the pressure/airflow, volume/lumen relation and its possible changes after mandibular repositioning and maxillary expansion in children will lead to a better understanding of how orthodontics could potentially affect the upper airway. Previous studies have reported a link between mandibular advancement appliances and maxillary appliances to an increase in the upper airway volume. However, more studies are needed to evaluate the relationship between the changes in the upper airway volume and actual airflow and respiratory capability. The airway volume measurement is important to, preliminary, state if there is an increase in the upper airway after orthodontic treatment.

However a change in shape, even with the same volume, can affect the pressure and airflow. In this sense, the pressure drop analysis will allow an answer to those questions

DETAILED DESCRIPTION:
Our hypotheses are:

1. There is an increase in upper airway volume and minimal cross-sectional area after maxillary expansion and mandible repositioning in class II malocclusion children using Hyrax and Twin-block.
2. There is a larger increase in the airway dimensions and a larger decrease in the air resistance (in the pressure drop analysis) in the group started with the mandibular advancement device.
3. There is a change in the shape of the upper airway after maxillary expansion and mandible repositioning in class II malocclusion children using Hyrax and Twin-block.
4. There is a correlation between the increase in airway volume, the change in shape and an increase in airflow using in vitro simulated airway experiments.
5. There is an increase in respiratory capability when evaluated with in-home portable PSG (after maxillary expansion and mandible repositioning).
6. There is a positive correlation to the in-home portable Polysomnography (PSG) with the results acquired by volume, shape, airflow and pressure drop.

Methods

The inclusion criteria are children between the ages 8-14 years old (8-12 years old girls and 9-14 years old boys), presenting skeletal class II division 1 malocclusion with maxillary constriction. The study design is a randomized crossover controlled trial. 90 patients will be randomly allocated into three groups:

Group 1: 30 patients will immediately undergo to Hyrax/Twin-block treatment, the patients will have the maxillary expansion treatment (Part I) before the mandibular repositioning (Part II).

Group 2: 30 patients will immediately undergo Twin-block/Hyrax treatment, the patients will have the mandibular repositioning treatment (Part I) done before the maxillary expansion (Part II).

Group 3: 30 patients will wait 1,5 years to begin the treatment. Since all patients are in the pre-pubertal/pubertal phase, this 1,5-year delay treatment for group 3 will neither compromise future treatment decisions nor results.

Aim 1: To determine the changes in the upper airway volume, minimal cross-sectional area, the lumen (geometry/shape), airflow, air velocity and pressure after maxillary expansion and mandibular advancement in children. Those changes will be compared between tested and control groups.

The upper airway will be assessed through Cone Bean Computed Tomography (CBCT)s exams, to analyze the volume changes before and after the use of the Twin-block and Hyrax, using the Avizo software (Thermo Fisher Scientific, Berlin, Germany). The pressure drop will be assessed using the CBCTs to generate a Stereolithography (STL) file to print upper airway models to analyze airflow, air velocity and pressure characteristics before and after the orthodontic treatment in children. Those results will be correlated. Also, the correlation will be done between tested and control groups. Pressure drop related measurements and airway volume will be assessed at T0 - before treatment, T1- after part II in the treated groups and T0 and after 1.5 years in the control group.

Aim 2: To determine changes in the in-home portable PSG results before and after maxillary expansion and mandibular repositioning and to correlate them to the results collected by the upper airway model's evaluations using pressure drop to determine airflow, velocity, pressure, and upper airway dimensions.

Patients will undergo an in-home PSG test at the beginning of treatment (T0). Groups 1 and 2 will have in-home PSG tested again after Part I and II. Group 3 will be tested at T0 and after one year. Through the CBCTs the volume and minimal cross-sectional area, and related measurements to pressure drop test will be assessed and correlated to the results from the in-home portable PSG. Likewise, the changes will be compared between tested and control groups.

Aim 3: To describe dental and skeletal changes in the class II patients undertaken the Twin-block/Hyrax treatment.

Linear measurements using craniofacial landmarks will be assessed through CBCT exams to determine the amount of skeletal and dental changes obtained. All patients will have those measurements assessed at T0. Groups 1 and 2 will also have linear measurements assessed after Part II. Group 3 will have linear measurements reassessed after 1.5 years from the first CBCT.

General information The CBCTs will be analyzed using Avizo software (Thermo Fisher Scientific, Berlin, Germany) for volume and linear measurement. Printed upper airway for the Pressure drop test for airflow/pressure drop/air velocity simulations will be made at all time-points.

All patients will have breathing capacity tested through in-home portable PSG, one week before the beginning of treatment, after parts I and II in groups 1 and 2 and at T0 and 1.5 years after the first test for group 3.

A subjective evaluation of the airway using the questionnaire Nasal Obstruction Symptom Evaluation (NOSE) Instrument, with 18 questions, will be given to patients. A Paediatric Sleep Questionnaire (PSQ) will also be used. An objective airway evaluation will be made using Peak Nasal Inspiratory Flow (PNIF) and Peak Oral Inspiratory Flow (POIF) tests, which are measured with the In-Check medical device at the same time-points as in-home PSG tests. Those tests and questionnaires will be used to correlate all the findings and clinical significance.

ELIGIBILITY:
Inclusion Criteria:

* children between the ages 8-14 years old (8-12 years old girls and 9-14 years old boys), presenting skeletal class II division 1 malocclusion with maxillary constriction

Exclusion Criteria:

* syndromic patients, previous ortho history, non-compliance, severe oral health issues (cavities, poor oral hygiene)

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Airflow | 3 years
  Airflow of the upper airway using pressure drop experimental analyzed using the CBCTs scans to print out the models of the upper airway.

SECONDARY OUTCOMES:
Dental changes | 3 years
  Dental changes after orthodontic treatment. Measurements of the teeth in relation to several cranial based landmarks will be made to analyse teeth movements. Those measurements will be done using the CBCTs scans.
Skeletal changes | 3 years
  Skeletal changes after orthodontic treatment. Measurements of 29 landmarks inside the skull will be made to verify the changes related to bone. The CBCTs scans will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia G Capenakas, MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Data won't be shared for confidential reasons and all data will be grouped.